CLINICAL TRIAL: NCT05566912
Title: AVOIDING PAIN CAUSED BY INSULIN INJECTION Patients Using Insulin With Diabetes Seek For Painless Injection
Brief Title: Practices Made by Patients to Avoid Insulin Injection Pain
Status: Completed | Type: Observational
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Halil Ibrahim Tuna PhD, Director, Selcuk University
Other Study IDs: Insulin Injection Pain
Record Dates: First submitted 2022-09-27; First posted 2022-10-05 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Diabetes Mellitus
Keywords: Insuline injection pain; lipohypertrophy; nursing care
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 7 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: filling out a survey — This research is a descriptive study

SUMMARY:
Abstract Objective: This study was conducted to determine the knowledge levels of DM patients about the disease and insulin use, and their practices to avoid insulin injection pain.

Methods: Data were collected from 399 patients who administered insulin injections in the study. Patient identification form, disease and treatment compliance form, Morisky-8 Treatment Adherence Scale (MMAS-8), and Visual Analog Scale were used for data collection. The data were collected by the same researcher by face-to-face interview technique.

DETAILED DESCRIPTION:
The face-to-face interview technique was applied to all patients who met the inclusion criteria and accepted to participate in the study, in the waiting area of the internal medicine outpatient clinic. Data were collected by the same researcher. Questionnaire forms were filled in the form of questions and answers in 10-15 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18-65, diagnosed with diabetes mellitus at least 1 year ago, injecting themselves with insulin.

Exclusion Criteria:

* Having no communication problems, and having no mental illness were included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with diabetes between the ages of 18-65
Sampling Method: Non-Probability Sample
Enrollment: 399 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Completing the surveys | 7 months
  Completion of all questionnaires by patients

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, Konya, Akşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No